CLINICAL TRIAL: NCT04483934
Title: Treatment of Patients With Non-healing Wounds and Trophic Ulcers Using Local LED Phototherapy and Autologous Dermal Fibroblasts
Brief Title: Treatment of Patients With Non-healing Wounds and Trophic Ulcers Using Autologous Dermal Fibroblasts
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Minsk Scientific-Practical Center for Surgery, Transplantation and Hematology (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_Fibr(TrophicUlcer)
Record Dates: First submitted 2020-07-17; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Trophic Ulcer; Non-healing Wound; Non-Healing Ulcer of Skin
Keywords: Trophic Ulcer; Non-healing Wound; Dermal fibroblasts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with dermal fibroblasts (Experimental): Cultured dermal fibroblasts and LED phototherepy
  Interventions: Biological: Dermal fibroblasts; Device: LED phototherapy

INTERVENTIONS:
Biological: Dermal fibroblasts — Cultured autologous dermal fibroblasts.
  For PR: The name "dermal fibroblasts" is exactly the name of the cell product registered by our ministry of health. There is no trade or international name.
Device: LED phototherapy — LED phototherapy

SUMMARY:
Treatment of patients with non-healing wounds and trophic ulcers using local LED phototherapy with local transplantation of autologous dermal fibroblasts

DETAILED DESCRIPTION:
During the implementation of the project, it was planned to develop a method for the treatment of trophic ulcers using injection of autologous dermal fibroblasts in the wound.

The positive outlook for the effectiveness of photodiode therapy with dermal fibroblasts is due to the following:

* the ability of fibroblasts to stimulate tissue regeneration
* positive results of preclinical studies of the method of treatment of long-term non-healing wounds in animals (rats).

Twelve patients were included in the study. Dermal fibroblasts were isolated from the skin patients, cultured and then transplanted back to the wound.

The therapeutic dose of cells was 50k per cm2 of the wound area. Follow up patients monitoring was performed at 1, 2 and more months after injection.

ELIGIBILITY:
Inclusion Criteria:

* Trophic Ulcers
* Chronic non-healing wounds

Exclusion Criteria:

* acute and chronic infectious diseases: HIV, viral hepatitis, tuberculosis
* mental disorders
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with tropic ulcers cured | 1 month
  Number of patients cured
Number of patients with treatment-related adverse events | 4 weeks
  Fibroblasts injection related adverse events assessed by blood count and function tests

CONTACTS AND LOCATIONS:
Overall Officials: Igor Volotovski, Prof, Study Director — Head of the Lab of Institute of Biophysics and Cell Engineering; Stanislav Tretyak, Prof, Study Director — Head of 2nd Department of Surgical Diseases of BSMU; Evgeny Baranov, Dr, Principal Investigator — Ass prof of 2nd Department of Surgical Diseases of BSMU; Zinaida Kvacheva, Dr, Principal Investigator — Lead Researcher of Institute of Biophysics and Cell Engineering
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No